CLINICAL TRIAL: NCT06632925
Title: Utility of Analyzing Atrial Signal Electrograms in Patients with Atrial Fibrillation Using Next-Generation Ensite X Software: a Prospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chin-Yu Lin, Taipei Veterans General Hospital, Department of Heart Rhythm Center and Cardiovascular Center. Associate Professor, School of Medicine, National Yang-Ming Chiao Tung University., Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2024-03-001A
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Ensite X Software; Atrial arrhythmia; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: Catheter ablation — The catheter ablation strategy is the same as the current treatment approach in patients with AF, according to the consensus of catheter ablation of AF. All procedures will be performed under local sedation or general anesthesia depending on the operator, and each patient will undergo an electrophysiological study and substrate mapping in the fasting state with adequate pre-ablation anticoagulation and transesophageal echocardiography to rule out LA thrombus. All antiarrhythmic drugs except amiodarone will be discontinued for at least 5 half-lives before the procedure.
  Step I: Substrate mapping before ablation, Step II: Pulmonary vein isolation (PVI), Step III: Post-ablation mapping in SR immediately after ablation, Step IV: Inducibility after ablation, Step V: Remmaping 30 minutes after ablation

SUMMARY:
A single-center clinical trial on the analysis of intracardiac atrial electrogram mapping before and after ablation with the HD Grid Mapping Catheter and Ensite X Software, as a prospective study.

DETAILED DESCRIPTION:
This study was designed to determine the efficacy of substrate ablation using HD Grid Mapping Catheter could collected more AF electrogram and facilitate the mapping resolution and driver identification in AF patients who required substrate modification. This study is a prospective, single-center in which patients with AF who will receive catheter ablation.

The priority of substrate modification would be determined by the mapping with the HD Grid mapping catheter. The end-point of ablation is non-inducible of AF or AFL. The procedure time, fluoroscopic time, procedural termination rate, and recurrence of atrial arrhythmia would be collected. If the flutter or the non-PV triggers were inducible, isthmus ablation and the non-PV trigger ablation will be performed accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Patents who sign the informed consent forms, and allow to be followed.
2. Symptomatic AF refractory or intolerant to at least one Class 1 or 3 antiarrhythmic medication.
3. Patients with age equal or greater than 20 years old regardless of gender.

Exclusion Criteria:

1. The presence of a atrial or ventricular thrombus.
2. Patients who are allergic to or unsuitable for use with the contrast media.
3. Pregnant patients or patients who are unavailable to receive X-ray.
4. Patients with renal insufficiency.
5. Patients had autonomic nervous system disorder (e.g. respiratory apnea)
6. Patients with age less than 20 years old or greater than 80 years old regardless of gender.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criteria for inclusion (same as current inclusion criteria for catheter ablation of
  AF):
  1. Patents who sign the informed consent forms, and allow to be followed.
  2. Symptomatic AF refractory or intolerant to at least one Class 1 or 3 antiarrhythmic medication.
  3. Patients with age equal or greater than 20 years old regardless of gender.
  Criteria for exclusion (same as current inclusion criteria for catheter ablation of
  AF):
  1. The presence of a atrial or ventricular thrombus.
  2. Patients who are allergic to or unsuitable for use with the contrast media.
  3. Pregnant patients or patients who are unavailable to receive X-ray.
  4. Patients with renal insufficiency.
  5. Patients had autonomic nervous system disorder (e.g. respiratory apnea)
  6. Patients with age less than 20 years old or greater than 80 years old regardless of gender.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Single-procedure freedom from AF | From the catheter ablation date to 12 months
  The study's primary endpoint was single-procedure freedom from AF after a blanking period based on a single procedure.
  After discharge, the patients were followed up (two weeks after the catheter ablation, then every 3 months) at our cardiology clinic or with the referring physician. During each follow-up, 24-hour Holter monitoring, or cardiac event recording was performed for a week. A 7-day holter will be performed in the 6th and 12th months. Recurrence was defined as any atrial arrhythmia recurrence, including AF and atrial tachycardia, and was defined as an episode lasting >1 minute and confirmed by ECGs months after the ablation.

SECONDARY OUTCOMES:
Non-inducibility of AF or AFL | During catheter ablation procedure
Any recurrence of all atrial arrhythmias after the first procedure | In the 6th and 12th months after catheter ablation.
  A 7-day holter will be performed in the 6th and 12th months.
Safety | From the catheter ablation date to 12 months follow-up
  This outcome measure will assess the procedural time, radiation exposure time, and the incidence of major complications, including cardiac tamponade, peripheral aneurysm, cerebral infarction, and shock

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided